CLINICAL TRIAL: NCT05469542
Title: Correlation of Electrocardiographic Signals Acquired by a Finger-worn ECG Sensor With a Standard 12-Lead ECG
Brief Title: Everbeat Ring ECG Clinical Concordance Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grektek Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00064656
Record Dates: First submitted 2022-07-04; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Diseases
Keywords: ECG; Wearables; Electrocardiography
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Everbeat Ring — The primary objective of this study is to assess the concordance of specific ECG parameters obtained in the everbeat nine-lead ECG waveform with those obtained in the comparable leads from a standard 12-lead ECG recorder.

SUMMARY:
This study is a cross-sectional observational study conducted in patients referred for routine ECG, to compare output from the everbeat finger-worn ECG device to standard of care (SOC) 12-lead electrocardiography. No intervention is involved in this study. Patients visiting the study site during the study period will be assessed for eligibility on a convenience basis, and observational data will be recorded on those eligible.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 90 years.
* Under the care of a board-certified physician and referred for a routine electrocardiogram (ECG)
* Resting heart rate between 50 to 120 beats per minute (BPM).

Exclusion Criteria:

* Inability to wear the everbeat ring.
* Prior history of movement disorders including Parkinson's or benign tremors.
* Prior history of allergic skin reactions to metal including stainless steel.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-90 presenting for a routine internal medicine or cardiology clinic visit
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-09-20 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
R-wave Amplitude | 50 days
  R Peak Amplitude intraclass correlation coefficient between test and reference devices in mm
ST-segment | 50 Days
  Concordance in ST-segment deviation from the TP segment if present in mm
Blinded Cardiologist Review | 50 Days
  Identify the first six consecutive distinct readable PQRST complexes without artifacts that match between the strips for evaluation. Each reviewer will assign a pass/fail to the strips by visually assessing all 6 PQRST complexes. A "pass" is given when the morphology of the PQRST complexes appears to overlay to the unaided eye. A measurement of the R amplitude from the isoelectric baseline to the nearest millimeter for the first two QRS complexes in both the reference strip and everbeat strip. The reviewers will be blinded to the identity of the reference strip and everbeat strip.

SECONDARY OUTCOMES:
User acceptance survey | 50 days
  To assess the ease of use of the everbeat ring in a random selection of users.

CONTACTS AND LOCATIONS:
Locations (1):
- BKLYNCardio, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided